CLINICAL TRIAL: NCT00489073
Title: Duloxetine Versus Placebo in the Treatment of Fibromyalgia Patients With or Without Major Depressive Disorder
Brief Title: Duloxetine Versus Placebo for Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6158; F1J-MC-HMCA
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2007-06-21 (Estimated); Status verified 2007-06

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: duloxetine
Drug: placebo

SUMMARY:
The primary purpose of this study is to determine if duloxetine reduces pain severity in patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* You are male or female outpatient at least 18 years of age with fibromyalgia. Females of child-bearing potential must test negative on a pregnancy test at visit 1.

Exclusion Criteria:

* Serious or unstable cardiovascular, hepatic, renal, respiratory, or hematologic illness, symptomatic peripheral vascular disease, or other medical condition (including unstable hypertension and not clinically euthyroid) or psychological conditions that in the opinion of the investigator would compromise participation or be likely to lead to hospitalization during the course of the study.
* Abnormal thyroid-stimulating hormone concentrations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345
Dates: Start 2002-11; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
To assess efficacy of duloxetine 60 mg twice daily (BID) compared with placebo on reduction of pain severity, measured by average pain item of Brief Pain Inventory (BPI) in patients with ACR-defined primary fibromyalgia, with or without major depression.

SECONDARY OUTCOMES:
To evaluate the efficacy of duloxetine 60 mg once daily (QD) compared with placebo during a 12-week, double-blind, acute therapy phase on the reduction of pain severity as measured by the average pain item of the Brief Pain Inventory (BPI).
To evaluate efficacy of duloxetine 60 mg QD and 60 mg BID vs. placebo during a 12-week, double-blind, acute therapy phase on the improvement of the area under the curve of pain relief as derived from BPI average pain score
To evaluate efficacy of duloxetine 60 mg QD and 60 mg BID vs. placebo during a 12-week, double-blind, acute therapy phase on the improvement of Fibromyalgia Impact Questionnaire (FIQ) total score
To evaluate efficacy of duloxetine 60 mg QD and 60 mg BID vs. placebo during a 12-week, double-blind, acute therapy phase on improvement of Brief Pain Inventory (BPI) severity (worst pain, least pain, pain right now) and interference scores
To evaluate efficacy of duloxetine 60 mg QD and 60 mg BID vs. placebo during a 12-week, double-blind, acute therapy phase on the improvement of Tender point pain thresholds: mean thresholds and number of points with a low threshold
To evaluate efficacy of duloxetine 60 mg QD and 60 mg BID vs. placebo during a 12-week, double-blind, acute therapy phase on the improvement of Clinical Global Impression of Severity (CGI)
To evaluate efficacy of duloxetine 60 mg QD and 60 mg BID vs. placebo during a 12-week, double-blind, acute therapy phase on the improvement of Patient Global Impression of Improvement (PGI)
To evaluate efficacy of duloxetine 60 mg QD and 60 mg BID vs. placebo during a 12-week, double-blind, acute therapy phase on the improvement of Hamilton Depression 17- item Rating Scale (HAMD17) total score
To demonstrate that the effect of duloxetine 60 mg QD and duloxetine 60 mg BID on the BPI average pain score is independent of the presence or absence of a major depressive disorder (MDD) as defined by DSM-IV.
To evaluate whether improvement in pain severity (assessed by BPI average pain score) is direct analgesic effect of duloxetine therapy and independent of treatment effect on mood improvement, as measured by total score of HAMD17

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com